CLINICAL TRIAL: NCT04672707
Title: Study on the Pharmacokinetics of Bromine Hexane Hydrochloride Tablets in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Wanbangde Pharmaceutical Group Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCYY-BEFA-2020BCCT002
Record Dates: First submitted 2020-12-13; First posted 2020-12-17 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Bromhexine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Bromhexine Hydrochloride Tablet, 32 mg, 8 mg 4 tablets, three times a day, for 2 days
  Interventions: Drug: Bromhexine Hydrochloride Tablet
- Group B (Experimental): Bromhexine Hydrochloride Tablet, 48 mg, 8 mg 6 tablets, three times a day, continuous service within 2 days
  Interventions: Drug: Bromhexine Hydrochloride Tablet
- Group C (Experimental): Bromhexine Hydrochloride Tablet, 64 mg ,8 mg spec 8 tablets ,3 times daily ,2 days in succession)
  Interventions: Drug: Bromhexine Hydrochloride Tablet
- Group D (Experimental): Bromhexine Hydrochloride Tablets, 80 mg ,8 mg Standard preparation 10 tablets ,3 times a day ,2 day
  Interventions: Drug: Bromhexine Hydrochloride Tablet

INTERVENTIONS:
Drug: Bromhexine Hydrochloride Tablet — 32 mg
  Arms: Group A
Drug: Bromhexine Hydrochloride Tablet — 48 mg
  Arms: Group B
Drug: Bromhexine Hydrochloride Tablet — 64 mg
  Arms: Group C
Drug: Bromhexine Hydrochloride Tablet — 80mg
  Arms: Group D

SUMMARY:
This clinical study is about increasing the dosage of bromine hexane hydrochloride to safety volume and continue to give it frequently in the new crown virus treatment could improve the efficacy.

DETAILED DESCRIPTION:
The purpose is to study the pharmacokinetic characteristics and safety of bromine hexane hydrochloride in healthy adults after oral administration of bromine hexane hydrochloride tablets. Then to explore the mechanism related to the role of transmembrane serine proteases (TMPRSSs) through the study, and to provide the basis for the clinical rational administration of bromine hexane hydrochloride tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and non-pregnant non-lactating females aged 18-55 years, including boundary values, trial period Over 55 years of age);
2. Male body weight ≥50 kg, female body weight ≥45 kg, body mass index (BMI )19,282 Between, including boundary values;
3. Health, no heart, liver, kidney, digestive tract, nervous system, mental disorders and metabolic disease history;
4. Sign informed consent before the trial, fully understand the content, process and possible adverse reactions, and communicate well with the researchers.

Exclusion Criteria:

1. Have participated in any clinical trial within 90 days before the trial or plan to participate in other clinical trials during the trial;
2. Have undergone major surgery within 90 days before the trial or plan to undergo surgery within 3 months after the trial;
3. Blood loss or donation of more than 300 blood mL (excluding female physiological blood loss) within 90 days prior to the trial, or blood transfusion;
4. Suffering from esophageal reflux, gastric bleeding or peptic ulcer disease within 180 days prior to the trial, more than once a week with heartburn, or any surgical procedure that may affect drug absorption (e.g. cholecystectomy);
5. a person with a specific history of allergies (asthma, urticaria, eczema, etc.), or an allergic constitution (e.g. allergic to two or more drugs, food or pollen), or a known component of the drug*or analogues/lactose allergy/intolerance;

   *The main components of the test drug: bromine hexane hydrochloride, excipients: starch, lactose, magnesium stearate.
6. Use of any medication within 28 days prior to the trial, including the use of prescription, over-the-counter and/or alternative medicines (e.g., medicinal meals, herbal medicines, hemostatic or health products) and the use of hormonal contraception or vaccines;
7. History of substance abuse;
8. Urine screening for substance abuse (tetrahydrocannabinol, benzodiazepine, barbiturates, morphine, cocaine, methamphetamine) was positive;
9. More than 3 cigarettes per day during the 90 days before the test; Alcoholism, Over 7 drinks per week for women and over 14 drinks per week for men (1=150 mL wine =360 mL beer and 45 spirits);
10. Positive breath test;
11. The body temperature (ear temperature)≥37.5℃, the respiration was obviously abnormal, and the researchers thought it was not suitable to take part in the experiment. The systolic blood pressure >140 mmHg or <90 mmHg, diastolic blood pressure (diastolic blood pressure) was 90 mmHg or 60 times 100/min or >;
12. Positive human immunodeficiency virus antibody (HIV-Ab), hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (HCV-Ab) or Treponema pallidum specific antibody (TPHA);
13. There are special requirements for diet, during the test can not comply with a unified diet;
14. Subjects refused to comply with the 48-hour ban on caffeine, alcohol, grapefruit and food (including tea, chocolate, coffee, cola, etc.);
15. Participants with partners refused to use effective contraception within 180 days from screening to completion of the trial；
16. Female subjects were positive for blood/urine pregnancy;
17. (c) Persons with renal insufficiency, impairment or previous urinary system disease;
18. hereditary galactose intolerance, lactase deficiency, or glucose-galactose malabsorption;
19. Halo acupuncture, halo blood and venous blood collection difficulties;
20. The physical examination has an obvious abnormality, and the researcher thinks it is not suitable to participate in the experiment;
21. Electrocardiogram examination has an obvious abnormality, and the researcher thinks it is not suitable to participate in the experiment;
22. Blood biochemistry, blood routine, urine routine examination have obvious abnormal, and the researchers think it is not suitable to participate in the test;
23. The subjects may not be able to complete the study for other reasons or may not be suitable for participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 48 hours
  Maximum observed concentration

SECONDARY OUTCOMES:
Area under curve (AUC 0-16h) | up to 48 hours
  16 hour dosing period; 3 dosing periods each separated by 2 day washout
AUC(AUC to infinity) | up to 48 hours
  16 hour dosing period; 3 dosing periods each separated by 2 day washout
AUC_%Extrap | up to 48 hours
  The proportion of the AUC (AUC to infinity) from the last point until we theoretically extrapolate to infinity
Time of maximum concentration (Tmax) | 2 to 2.5 hours
  16 hour dosing period; 3 dosing periods each separated by 2 day washout
Clearance rate（CL） | up to 48 hours
  Apparent clearance rate
Vd | up to 48 hours
  Apparent volume of distribution
t1/2 | 5 hour
  16 hour dosing period; 3 dosing periods each separated by 2 day washout
λz | up to 48 hours
  Terminal disposition rate constant

CONTACTS AND LOCATIONS:
Locations (1):
- The 2nd Second Affiliated Hospital of WMU Phase I Clinical Trial Unit /Center Of Bioequivalence Study, Wenzhou, Zhejiang, China